CLINICAL TRIAL: NCT06421753
Title: Efficiency of Spatially Distributed Sequential Stimulation (Sdss) for Functional Electrical Stimulation (FES) of Upper Motor Neuron Syndrome (UMR) Patients
Acronym: SDSS_UMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UGECAM Rhône-Alpes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-01-VR
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-05

CONDITIONS: Upper Motor Neuron Disease
Keywords: functional electrical stimulation; muscle fatigue; rehabilitation; spinal cord injury; stroke; multiple sclerosis
MeSH Terms: conditions — Motor Neuron Disease; Spinal Cord Injuries; Stroke; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: SCED : Single Case Experimental Design Each patient is his own control Patient will be randomised to receive FES-cycling with SDSS or standard electrical stimulation
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spatially Distributed Sequential Functional Electrical Stimulation (Experimental): Interventions: 3 FES cycling sessions separated by 48h of rest. Each session is comprised of 2 phases separated by 20 minutes of rest. Each phase is comprised of a 3 minutes passive cycling warm-up, followed by 3 minutes of electrically stimulated cycling.
  Interventions: Device: SDSS
- Standard Electrical Stimulation During Functional Electrical Stimulation (Active Comparator): Each session begins with a 3-minute warm-up phase, followed by a 3-minute stimulation phase. The motor rotates the legs at 50 rpm during both phases. The type of stimulation used in the first phase is chosen randomly. After a 20-minute break, the second warm-up and stimulation phases are carried out. During the second session, the order of the stimulation phases is reversed.
  Interventions: Device: Standard Electrical Stimulation During Functional Electrical Stimulation

INTERVENTIONS:
Device: SDSS — Each session begins with a 3-minute warm-up phase, followed by a 3-minute stimulation phase. The motor rotates the legs at 50 rpm during both phases. The type of stimulation used in the first phase is chosen randomly. After a 20-minute break, the second warm-up and stimulation phases are carried out During the second session, the order of the stimulation phases is reversed.
  Arms: Spatially Distributed Sequential Functional Electrical Stimulation
Device: Standard Electrical Stimulation During Functional Electrical Stimulation — Each session begins with a 3-minute warm-up phase, followed by a 3-minute stimulation phase. The motor rotates the legs at 50 rpm during both phases. The type of stimulation used in the first phase is chosen randomly. After a 20-minute break, the second warm-up and stimulation phases are carried out During the second session, the order of the stimulation phases is reversed.
  Arms: Standard Electrical Stimulation During Functional Electrical Stimulation

SUMMARY:
To determine whether Spatially Distributed Sequential Functional Electrical Stimulation is more effective than Standard Electrical Stimulation During Functional Electrical Stimulation in Upper Motor Neuron Patients

DETAILED DESCRIPTION:
Design: SCED (single case experimental design) prospective, monocentric, comparative interventional study (SDSS versus SES) Population: patients with motor deficit due to upper motor neuron syndrome Setting: Neurologic Rehabilitation Unit Interventions: 3 FES cycling sessions separated by 48h of rest. Each session is comprised of 2 phases separated by 20 minutes of rest. Each phase is comprised of a 3 minutes passive cycling warm-up, followed by 3 minutes of electrically stimulated cycling.

Participants will be evaluated before and during the training.

ELIGIBILITY:
Inclusion Criteria:

Patients with Upper Motor Neuron syndrome:

* adult (> 18 years)
* motor deficit due to an acquired traumatic or neurodegenerative motor deficiency of the central nervous system (MRC<4/5)
* stable clinical condition, particularly on the cardiovascular level (recent assessment by a cardiologist with stress test)
* non denervated muscles
* tolerant to muscle electrical stimulation
* having given written consent
* able to cycle 30 minutes with FES-cycling

Exclusion Criteria:

* major cognitive comprehension disorders that could compromise understanding of the protocol and the smooth running of the study
* cardiac pacemaker and other contraindications relating to the use of electrostimulation (in particularly "deep vein thrombosis")
* spasticity of the lower limbs making flexion/extension movement difficult
* participation in another study
* pregnancy
* people with the following legal and administrative states or situations:
* people placed under judicial protection;
* persons deprived of their liberty, persons subject to psychiatric care and persons admitted to a health or social establishment for purposes other than that of clinical investigation;
* unemancipated minors;
* people who are not affiliated to a social security scheme or beneficiaries of such a scheme

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Average quadriceps power output (watts) measured during 3 minutes of FES cycling | during sessions of FES cycling
  The subjects are installed on a Hepha Bike electrostimulation bike, equipped with force-torque measuring pedals (ICS_RM, Sensix, France), synchronized with a MotiMove-8 stimulator. The average quadriceps power (watts) during the first and last 30 seconds of each stimulation phase, as well as the total average power (Pm) are calculated.

SECONDARY OUTCOMES:
Evaluate the comfort of dry and hydrogel based functional electrical stimulation electrodes | before the first session of FES cycling
  Dry electrode then hydrogel electrode are placed on the quadriceps' motor point The amplitude of stimulation is increased in steps of 3 mA followed by 5 seconds of rest for subsequent trains until the subject feels a burning sensation. the stimulation threshold (mA) is compared between dry and hydrogel electrode

CONTACTS AND LOCATIONS:
Locations (1):
- SMR Val Rosay, Saint-Didier-au-Mont-d'Or, France, France

IPD SHARING:
Plan to Share IPD: No